CLINICAL TRIAL: NCT03341286
Title: Randomized, Placebo Controlled, Phase II Trial, on the Effect of an Oral Supplement,TK3 (Tryptophan and Thiamine) on the Quality of Life and Chemotherapy Tolerance in Cancer Patients With Advanced Disease.
Brief Title: The Effect of an Oral Supplement,TK3 (Tryptophan and Thiamine) on the Quality of Life and Chemotherapy Tolerance in Cancer Patients With Advanced Disease.
Acronym: TK3bFIIABC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Daniel de Iracema Gomes Cubero, PHD, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TK3b FII ABC
Record Dates: First submitted 2017-09-22; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Cancer; Quality of Life; Chemotherapy Effect; Tryptophan; Thiamine
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TK3 (Experimental): This is a oral supplement combination of tryptophan and thiamine called TK3 to be taken three times a day
  Interventions: Drug: TK3
- Placebo (Placebo Comparator): Placebo orally, to be taken three times a day
  Interventions: Drug: TK3

INTERVENTIONS:
Drug: TK3 — Tryptophan and thiamine as on oral supplement

SUMMARY:
The product under investigation relates to a pharmaceutical composition containing a pyrimidine nitrogen base, thymine, and the essential amino acid tryptophan. This product seems to have effect on quality of life and enhance adverse affects of chemotherapy in cancer patients.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the impact of TK3 on the quality of life of patients receiving anti-neoplastic chemotherapy. The secondary objectives are to evaluate the influence of TK3 on the side effects caused by anti-neoplastic chemotherapy, tolerance to this treatment and the safety of the use of the TK3 product in cancer patients, accompanying the appearance of non-characteristic effects of the existing cancer type .

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to study procedures and sign the informed consent
* Patients 18 years of age or older;
* Patients undergoing oncologic treatment for advanced neoplasms. It is understood by advanced patient disease patients with unresectable or with distant metastases.
* Participants should present at least one (1) of the following clinical side effects that can be assessed according to CTCAE (Version 4.0): fatigue, nausea, vomiting, diarrhea, or mucositis.
* Patients with programming to receive at least 3 cycles of anti-neoplastic chemotherapy;
* Patients may be on radiotherapy

Exclusion Criteria:

* Use of vitamin complex or concomitant food supplement;
* Current use or programming of parenteral diet use;
* Hypersensitivity to the components of the formula;
* Participation in another clinical study or use of any investigational product within 28 days prior to commencement of treatment in this clinical trial, unless the Investigator deems there to be a clinical benefit therefore;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
The role of TK3 in the quality of life of patients receiving anti-neoplastic chemotherapy after 3 cicles of chemotherapy | It depends on the chemotherapy schedule: 14 or 21 days
  use of quality of life questionaire QLQ-C30
The role of TK3 in the quality of life of patients receiving anti-neoplastic chemotherapy after 3 cicles of chemotherapy | It depends on the chemotherapy schedule: 14 or 21 days
  use of quality of life questionaire FACIT-F

SECONDARY OUTCOMES:
The effects of TK3 on tolerance to anti-neoplastic chemotherapy, with emphasis on the most prevalent side effects, especially fatigue related to cancer treatment according to CTCAE scale of adverse events v 4.0 | It depends on the chemotherapy schedule: 14 or 21 days
  use of CTCAE scale of adverse events v 4.0 and Edmonton scale
Drugs safety according to CTCAE scale of adverse events v 4.0 | It depends on the chemotherapy schedule: 14 or 21 days
  safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de medicina do ABC-CEPHO, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Butt Z, Lai JS, Rao D, Heinemann AW, Bill A, Cella D. Measurement of fatigue in cancer, stroke, and HIV using the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) scale. J Psychosom Res. 2013 Jan;74(1):64-8. doi: 10.1016/j.jpsychores.2012.10.011. Epub 2012 Nov 15. PMID 23272990
- [Background] Watanabe SM, Nekolaichuk C, Beaumont C, Johnson L, Myers J, Strasser F. A multicenter study comparing two numerical versions of the Edmonton Symptom Assessment System in palliative care patients. J Pain Symptom Manage. 2011 Feb;41(2):456-68. doi: 10.1016/j.jpainsymman.2010.04.020. Epub 2010 Sep 15. PMID 20832987
- [Background] Bruera E, Kuehn N, Miller MJ, Selmser P, Macmillan K. The Edmonton Symptom Assessment System (ESAS): a simple method for the assessment of palliative care patients. J Palliat Care. 1991 Summer;7(2):6-9. PMID 1714502
- [Background] Monteiro Dda R, Almeida Mde A, Kruse MH. [Translation and cross-cultural adaptation of the Edmonton Symptom Assessment System for use in Palliative Care]. Rev Gaucha Enferm. 2013 Jun;34(2):163-71. doi: 10.1590/s1983-14472013000200021. Portuguese. PMID 24015476
- [Background] Cocks K, King MT, Velikova G, Martyn St-James M, Fayers PM, Brown JM. Evidence-based guidelines for determination of sample size and interpretation of the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30. J Clin Oncol. 2011 Jan 1;29(1):89-96. doi: 10.1200/JCO.2010.28.0107. Epub 2010 Nov 22. PMID 21098316
- [Background] Osoba D, Slamon DJ, Burchmore M, Murphy M. Effects on quality of life of combined trastuzumab and chemotherapy in women with metastatic breast cancer. J Clin Oncol. 2002 Jul 15;20(14):3106-13. doi: 10.1200/JCO.2002.03.090. PMID 12118024
- [Background] Cortes J, Hudgens S, Twelves C, Perez EA, Awada A, Yelle L, McCutcheon S, Kaufman PA, Forsythe A, Velikova G. Health-related quality of life in patients with locally advanced or metastatic breast cancer treated with eribulin mesylate or capecitabine in an open-label randomized phase 3 trial. Breast Cancer Res Treat. 2015 Dec;154(3):509-20. doi: 10.1007/s10549-015-3633-7. Epub 2015 Nov 14. PMID 26567010
- [Background] Curran D, Pozzo C, Zaluski J, Dank M, Barone C, Valvere V, Yalcin S, Peschel C, Wenczl M, Goker E, Bugat R. Quality of life of palliative chemotherapy naive patients with advanced adenocarcinoma of the stomach or esophagogastric junction treated with irinotecan combined with 5-fluorouracil and folinic acid: results of a randomised phase III trial. Qual Life Res. 2009 Sep;18(7):853-61. doi: 10.1007/s11136-009-9493-z. Epub 2009 Jul 1. PMID 19568958
- [Background] Brown J, Thorpe H, Napp V, Fairlamb DJ, Gower NH, Milroy R, Parmar MK, Rudd RM, Spiro SG, Stephens RJ, Waller D, West P, Peake MD. Assessment of quality of life in the supportive care setting of the big lung trial in non-small-cell lung cancer. J Clin Oncol. 2005 Oct 20;23(30):7417-27. doi: 10.1200/JCO.2005.09.158. Epub 2005 Sep 12. PMID 16157935
- [Background] Southwest Oncology Group; Berry DL, Moinpour CM, Jiang CS, Ankerst DP, Petrylak DP, Vinson LV, Lara PN, Jones S, Taplin ME, Burch PA, Hussain MH, Crawford ED. Quality of life and pain in advanced stage prostate cancer: results of a Southwest Oncology Group randomized trial comparing docetaxel and estramustine to mitoxantrone and prednisone. J Clin Oncol. 2006 Jun 20;24(18):2828-35. doi: 10.1200/JCO.2005.04.8207. PMID 16782921